CLINICAL TRIAL: NCT03549962
Title: Obesity is a Predictor of In-hospital Postoperative Complications in Patients Undergoing Elective Total Knee Arthroplasty
Brief Title: Preoperative Nutritional Status in Patients Undergoing Elective Total Knee Arthroplasty and In-hospital Postoperative Complications
Acronym: NUTR TKA
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Department of Orthopaedics & Traumatology; Director of MSc/PgD Programme in Musculoskeletal Medicine & Rehabilitation, Chinese University of Hong Kong
Other Study IDs: CUHK_2018.242
Record Dates: First submitted 2018-05-27; First posted 2018-06-08 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Preoperative Period; Nutritional Status; Arthroplasty Knee
Keywords: Preoperative; Nutritional Status; Arthroplasty; Replacement; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TKA — Total Knee Arthroplasty

SUMMARY:
Malnutrition has long been linked to postoperative complications and adverse outcomes in a variety of surgical fields , such as increased susceptibility to infection, delayed wound healing, and increased frequency of decubitus ulcers. In particular, it is a modifiable risk factor, as evident by studies that have associated optimization of preoperative nutrition with improved surgical outcomes. Therefore, it is important to identify these patients who are at risk so that appropriate nutritional support can be implemented.

A range of options for nutritional status assessment have been proposed; a comprehensive assessment may include measurements of dietary intake, clinical assessment, anthropometric measurements, and biochemical measurements of serum protein, micronutrients and metabolic parameters . Many of the signs of malnutrition, however, only manifest in extreme cases. Thus it is crucial to identify sensitive markers that can be utilized to screen for clinical as well as subclinical malnutrition patients.

In orthopaedic patients, the prevalence of clinical and subclinical malnutrition has been reported to be up to 42.4%. Common markers of malnutrition that have been studied include low serum albumin as a marker of protein status, low total lymphocyte count (TLC), and excessively high or low body mass index (BMI). They have been compared against various adverse surgical outcomes, including surgical site infections (SSI), delayed wound healing, unplanned intubation and ICU admission , postoperative anemia and cardiac complications , and length of hospital stay. However, conflicting results have been reported; for example, while hypoalbuminemia (serum albumin <3.5mg/dL) have been associated with increased risk of SSI and longer than average hospital stay, its effect on wound healing is less clear - Marin et al. reported no significant predictive value of hypoalbuminemia on wound healing, yet Greene et al. reported a 5-time increase in frequency of major wound complication.

The purpose of this retrospective cohort study was to identify biomarkers of malnutrition in patients undergoing elective total knee arthroplasty (TKA) that are predictive of adverse in-hospital postoperative complications, which would facilitate the identification of at risk patients for nutritional optimization before surgery.

Six-hundred and twenty-six patients who underwent elective TKA between 2013 and 2017 in the Prince of Wales Hospital in Hong Kong were reviewed; the preoperative serum albumin, TLC, and BMI were compared against in-hospital postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* All elective Total Knee Arthroplasty cases from 2013 to 2017
* All patients must have undergone elective Total Knee Arthroplasty in Prince of Wales Hospital Hong Kong

Exclusion Criteria:

* Revision of Total Knee Arthroplasty

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All elective Total Knee Arthroplasty cases from 2013 to 2017undergone elective Total Knee Arthroplasty in Prince of Wales Hospital Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 626 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
In-hospital postoperative complications | From March 2013 to December 2017
  deep surgical site or implant infection, hematoma requiring drainage, wound complications, systemic infection with identifiable source, unplanned intensive care unit (ICU) admission, deep vein thrombosis (DVT), pulmonary embolism (PE), neurological complications, acute renal failure, and cardiovascular complications

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Department of Orthopaedics & Traumatology, The Chinese University of Hong Kong, Hong Kong
  - Department of Orthopaedics & Traumatology, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided